CLINICAL TRIAL: NCT06533657
Title: A Phase 2A Study to Investigate the Safety and Preliminary Analgesic Efficacy of Oral Trichomylin® in Male and Female Participants 18 Years of Age and Above With Advanced Cancer and Moderate to Severe Cancer-Related Pain
Brief Title: Unique Treatment of Oncology Pain in Advanced Cancer
Acronym: UTOPIA-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ZYUS Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Z-TRI-10002A
Record Dates: First submitted 2024-07-25; First posted 2024-08-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cancer Pain
Keywords: Cannabinoid; Safety and Tolerability; Preliminary Efficacy; Opioid-sparing
MeSH Terms: conditions — Cancer Pain | interventions — Dronabinol; Cannabidiol; cannabichromene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trichomylin® (Experimental): Trichomylin® capsule (5 mg delta-9-tetrahydrocannabinol: 5 mg cannabidiol: 5 mg cannabichromene)
  Interventions: Drug: Trichomylin® capsule (5 mg delta-9-tetrahydrocannabinol: 5 mg cannabidiol: 5 mg cannabichromene)

INTERVENTIONS:
Drug: Trichomylin® capsule (5 mg delta-9-tetrahydrocannabinol: 5 mg cannabidiol: 5 mg cannabichromene) — Cancer patients meeting eligibility criteria will receive Trichomylin® and self-titrate to effective dose.

SUMMARY:
This will be a proof-of-concept, single arm study with a maximum of 20 patients to evaluate preliminary analgesic efficacy and safety of Trichomylin® in patients with advanced cancer (male and female) who suffer from moderate to severe chronic pain and who are taking a stable dose of long-acting opioid therapy for at least 1 week prior to screening.

DETAILED DESCRIPTION:
This study will consist of a screening visit, treatment, and safety follow-up period. There will be an initial patient determined titration phase, using escalated doses of Investigational Product, to reach a dose that achieves symptom relief with tolerable side effects. Each capsule of Trichomylin® contains a fixed ratio of 5 mg delta-9-tetrahydrocannabinol: 5 mg cannabidiol: 5 mg cannabichromene. Participants can titrate up to a maximum of 2 capsules twice daily (total of 4 capsules). This will be followed by a 5 day assessment period of the stable dose determined in collaboration with clinicians.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has voluntarily agreed to study participation by giving written informed consent and must be ≥18 years of age on the day of signing the informed consent form (ICF).
2. Participant has advanced solid malignant tumors not amenable to curative-intent therapy (locally advanced unresectable or metastatic).
3. Participant life expectancy is ≥3 months at screening according to investigator's best judgement.
4. Participant has a clinical diagnosis of moderate to severe cancer-related pain with average daily pain score to be ≥4 for at least 4 out of the 7-day screening period, despite ongoing opioid treatment, as evidenced by their response to the BPI-SF Question #5 on the Numeric Rating Scale (NRS).
5. Participant is taking a stable dose of opioid therapy (Step III according to the World Health Organization [WHO] analgesic ladder) for at least 1 week prior to screening to relieve cancer-related pain.
6. Participant has adequate organ function, as indicated by the following laboratory values, at screening:

   1. Baseline serum electrolytes must be within the normal range per local laboratories (for baseline serum electrolytes that are out of range, these may be corrected, and the potential participant may be rescreened).
   2. Stable renal function (estimated glomerular filtration rate [eGFR] >15).
   3. Total bilirubin (TBIL) ≤1.5 x upper limit of normal (ULN); or ≤3 x ULN for participants with Gilbert's syndrome.
   4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 x ULN or ≤5 x ULN for participants with liver metastases.
7. Participant has stable cardiac function, as determined by:

   1. No clinically significant ECG waveform abnormalities.
   2. QT interval corrected for heart rate using Fridericia's formula (QTcF) ≤470 msec, as determined by the mean QTcF values from the ECG assessments at screening (one triplicate).
8. Participant can tolerate oral medications including capsules.
9. Participant is willing to take a medication which may exhibit psychoactive effects.
10. Participant must discontinue the use of the following medications 7 days before the start of study intervention and for the duration of the trial, unless in the opinion of the investigator and sponsor, the medication will not interfere with the study: herbal supplements or related products which are cytochrome P450 (CYP) 2E1, CYP3A4, or P-glycoprotein substrates, or which are strong inhibitors of the CYP3A4 and/or CYP3A5 pathways or which are known CYP3A4 inducers (this includes grapefruit and Seville oranges juice or related products, and St. John's wort).
11. Participant must not engage in medicinal or recreational use of any cannabinoid containing substance, in any form, within 30 days prior to screening and be willing to abstain from medicinal or recreational use of cannabis and other cannabinoid compounds (other than the Investigational Product) for the duration of the study.
12. Participant must have a negative urine drug screen for cannabinoids at screening and prior to dosing at Day 1; one repeat test may be conducted for a suspected false positive result.
13. Participant must not have any current or past allergic or adverse reaction or known sensitivity to olive oil, gelatine, glycerin, and titanium dioxide, or to cannabinoid-like substances (including but not limited to dronabinol, marinol, nabilone, marijuana, cannabis, THC, or cannabinoid oil).
14. Female participants are eligible to enter and participate in the study if they are of:

    1. Non-childbearing potential.
    2. Childbearing potential with a negative serum pregnancy test at screening (within 7 days of the first dose of Investigational Product) and agree to use contraception before study entry and throughout the study until 3 months after the last administered dose of the Investigational Product.
15. Male participants are eligible to enter and participate in the study if they are vasectomized or agree to the use of contraception during the study treatment period and for at least 3 months after the last administered dose of the Investigational Product.
16. Participants, in the opinion of the investigator, should understand the nature of the study, be able to participate in all planned assessments, complete all required tests, and be likely to comply with all study procedures.

Exclusion Criteria:

1. Female participants who are pregnant or lactating.
2. Participant has uncontrolled psychiatric disorders (severe depression or anxiety, personality disorder, psychosis, or schizophrenia).
3. Participant has a family history of schizophrenia.
4. Participant has current or history of suicidal behavior or ideation assessed by Columbia-Suicide Severity Rating Scale (C-SSRS).
5. Participant has any known or suspected history of a diagnosed dependency disorder, including opioid abuse, current heavy alcohol consumption (i.e. more than 10 units of alcohol per week or 4 units on any given day [1 unit = 150 mL of wine, 260 mL of beer, or 45 mL of 40% alcohol]), current use of an illicit drug or current non-prescribed use of any prescription drug (Alcohol, Smoking and Substance Involvement Screening Test [ASSIST]).
6. Participant has engaged in medicinal or recreational use of any cannabinoid containing substance, in any form within the 30 days prior to screening.
7. Participant is within the first cycle of a new line of anticancer therapy (including but not limited to chemotherapy or other systemic anticancer therapies, immunotherapy, radiation therapy, or surgery) at the start of the screening period.
8. Participant has had any major surgery within 4 weeks prior to screening.
9. Participant has an active infection requiring systemic treatment at the start of the study treatment.
10. Participant has cirrhosis or severe hepatic impairment defined as AST and ALT >3 x ULN or >5 x ULN for participants with liver metastases.
11. Participant has any of the following cardiovascular criteria:

    a. Current evidence of unstable angina or another form of symptomatic cardiac ischemia b. Acute myocardial infarction ≤3 months prior to screening c. Heart failure of New York Heart Association Classification III or IV ≤3 months prior to screening d. Grade ≥2 ventricular arrhythmia ≤3 months prior to screening e. Cerebrovascular Accident (CVA) or Grade ≥2 Transient Ischemic Attack (TIA) ≤6 months prior to screening f. Grade ≥2 hypertension that cannot be managed by standard anti-hypertension medications before initiation of treatment g. Syncope or seizure ≤3 months before screening.
12. Participant has a history or presence of gastrointestinal disease or other condition known to interfere with the absorption of drugs.
13. Participant has intractable vomiting.
14. Participant has any other condition or abnormality that, in the investigator's judgement after medical interview, physical examination, and/or screening and baseline investigations, renders participant unfit for the study or precludes the participant's safe participation in and completion of the study.
15. Participant has concurrent participation in another therapeutic clinical trial or participation in another clinical trial within 30 days prior to the enrolment in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants That Reach the Stable Dose during Dose Titration | Baseline (i.e. Day 1 Dose Titration) and Stable Dose Day 1, up to 14 days
  Investigational Product will be titrated up incrementally until participants achieve their "optimal dose" that achieves symptom relief with tolerable side effects or to a maximum of 2 capsules twice daily. Once participants have had 2 full days (at minimum) of treatment at this dosage, this will then be considered their "stable dose".
Change in Average Pain Scores from Baseline to Investigational Product Discontinuation | Baseline and Investigational Product Discontinuation, up to 23 days
  The Brief Pain Inventory Short Form (BPI-SF) is a standardized scale used for capturing participant reported symptom assessments related to pain severity and the resulting functional interference caused by pain. The BPI-SF has a numerical rating scale used by participants to indicate their level of pain. Participants are asked to assign a number that best describes their pain on average from 0 = no pain, to 10 = pain as bad as you can imagine, at the same time every day during the Screening period (Day -7 to Day -1) and enter this number in response to the BPI-SF Question #5 on the evaluation form.
Proportion of Responders to Average Pain from Baseline to Investigational Product Discontinuation | Baseline and Investigational Product Discontinuation, up to 23 days
  Average pain as entered in response to the BPI-SF Question #5, where response is defined as having a baseline of ≥30% from baseline at the Investigational Product discontinuation visit.
Number of Participants That Reach the Stable Dose during Dose Titration and Respond to Average Pain from Baseline to Investigational Product Discontinuation | Baseline and Investigational Product Discontinuation, up to 23 days
  Participants have reached their "stable dose" and respond to average pain as entered in response to the BPI-SF Question #5, where response is defined as having a baseline of ≥30% from baseline at the Investigational Product discontinuation visit.
Change in Average Pain from Baseline to End of the Titration | Baseline and End of Dose Titration, up to 14 days
  Average pain as entered in response to the BPI-SF Question #5.
Change in Pain Interference from Baseline to End of the Titration | Baseline and End of DoseTitration, up to 14 days
  Pain interference is scored as the mean of the seven interference items and entered in response to the BPI-SF Question #9.
Change in Pain Interference from Baseline to Investigational Product Discontinuation | Baseline and Investigational Product Discontinuation, up to 23 days
  Pain interference as entered in response to the BPI-SF Question #9.

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | Baseline and End of Safety Follow-Up, up to 56 days
  The severity of an adverse events (AE) is graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 (NCI 2017). The incidence of AEs will be presented as the number (percentage) of participants with treatment emergent adverse events (TEAEs) by system organ class and Preferred Term using the most current Medical Dictionary for Regulatory Activities (MedDRA) available at the time of study commencement.
Incidence of Serious Adverse Events | Baseline and End of Safety Follow-Up, up to 56 days
  The incidence of serious adverse events (SAE) will be presented as the number (percentage) of participants with SAEs by system organ class and Preferred Term using the most current Medical Dictionary for Regulatory Activities (MedDRA) available at the time of study commencement.
Incidence of Adverse Events of Special Interest | Baseline and End of Safety Follow-Up, up to 56 days
  The incidence of adverse events of special interest (AESI) will be presented as the number (percentage) of participants with AESIs by system organ class and Preferred Term using the most current Medical Dictionary for Regulatory Activities (MedDRA) available at the time of study commencement.
Incidence of Adverse Events leading to Discontinuation of Study Treatment | Baseline and End of Safety Follow-Up, up to 56 days
  The incidence of adverse events (AE) leading to discontinuation of study treatment will be presented as the number (percentage) of participants with AEs by system organ class and Preferred Term using the most current Medical Dictionary for Regulatory Activities (MedDRA) available at the time of study commencement.
Change in Electrocardiogram From Baseline to Investigational Product Discontinuation | Baseline and Investigational Product Discontinuation, up to 23 days
  A triplicate 12-lead electrocardiogram (ECG) will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and [QTc] intervals.
Change in Brief Pain Inventory Short Form from Baseline to Investigational Product Discontinuation | Baseline and Investigational Product Discontinuation, up to 23 days
  The BPI-SF is a standardized scale used for capturing participant reported symptom assessments related to pain severity and the resulting functional interference caused by pain. The BPI-SF has a numerical rating scale used by participants to indicate their level of pain.
Proportion of responders in Brief Pain Inventory Short Form from Baseline to Investigational Product Discontinuation | Baseline and Investigational Product Discontinuation, up to 23 days
  The BPI-SF is a standardized scale used for capturing participant reported symptom assessments related to pain severity and the resulting functional interference caused by pain. The BPI-SF has a numerical rating scale used by participants to indicate their level of pain. Response is defined as having a decrease in pain from baseline by ≥30% at the Investigational Product discontinuation visit.
Change in Depression, Anxiety and Stress Scale - 21 Items from Baseline to Investigational Product Discontinuation | Baseline and Investigational Product Discontinuation, up to 23 days
  The Depression, Anxiety and Stress Scale- 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. By examining these subscales separately, DASS-21 provides a comprehensive picture of an individual's emotional state, aiding therapists, and researchers in identifying the primary areas of concern.
Change in Quality of Life and Functional Status from Baseline to Investigational Product Discontinuation | Baseline and Investigational Product Discontinuation, up to 23 days
  The European Organization for Research and Treatment of Cancer core Quality of Life (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological, and social functions. The questionnaire is composed of multi-item scales and single items (Version 3.0).
Change in Subjective Measures of Symptom Change from Baseline to Investigational Product Discontinuation | Baseline and Investigational Product Discontinuation, up to 23 days
  The Patient Global Impression of Change (PGIC) is a subjective measure of symptom change. Participants rate their change on a 7-point scale that ranges from "very much improved" to "very much worse", with "no-change" as the mid-point.
Use of Oral Morphine Equivalents from Baseline to Investigational Product Discontinuation | Baseline and Investigational Product Discontinuation, up to 23 days
  Rescue analgesia requirements, specifically use of opioid medications, both prescription and over the counter (OTC), will be documented at baseline and for the duration of the study. Opioid medications will be converted to morphine equivalent doses (MEDD) for comparison and evaluation purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Stakiw, MD, Study Director — Saskatoon Cancer Centre
Locations (3):
- Canada (3):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No